CLINICAL TRIAL: NCT01236885
Title: Use of a Computer-Guided Glucose Management System for Patients Undergoing Blood and Marrow Transplants (BMT)
Brief Title: Computer-Guided Glucose Management Systems in Treating Patients With Hyperglycemia Who Have Undergone Blood and Bone Marrow Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2425.00; NCI-2010-01102 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2425.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2010-11-04; First posted 2010-11-09 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Hyperglycemia; Malignant Neoplasm
MeSH Terms: conditions — Hyperglycemia; Neoplasms

ARMS (1):
- Supportive care (Glucommander) (Experimental): Patients receive blood glucose management with IV insulin using Glucommander.
  Interventions: Other: computer-assisted intervention

INTERVENTIONS:
Other: computer-assisted intervention — Undergo blood glucose management using Glucommander

SUMMARY:
This clinical trial studies computer-guided glucose management systems in treating patients with hyperglycemia who have undergone blood and bone marrow transplant. A computer-guided glucose management system may help manage glucose levels in patients who have undergone blood or bone marrow transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the ability of computer-guided glucose management system (CGGMS) algorithms to control glucose within or close to current University of Washington Medical Center (UWMC) intensive care unit (ICU) targets (100 to 140 mg/dl) in non-critically ill bone marrow transplant (BMT) adult (age >= 18 years) patients.

OUTLINE:

Patients receive blood glucose management with intravenous (IV) insulin using Glucommander.

ELIGIBILITY:
Inclusion Criteria:

* Post-transplant adult patients (age >= 18 years) on the BMT Service at UWMC
* Requiring insulin secondary to:

  * Known history of (h/o) type 2 diabetes mellitus
  * Two blood sugar values > 180 (point of care and/or am lab glycemia)
  * One blood sugar value > 250 (point of care or AM lab glycemia)

Exclusion Criteria:

* Critically ill patients (intensive care unit [ICU] admissions)
* Terminally ill patients
* Eastern Cooperative Oncology Group (ECOG) performance status > 3
* Previous type 1 diabetes mellitus
* Cognitively impaired patients, unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-12; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Percentage of glucose values within target range (100-140) by using CGGMS | Up to 2 years
  Standard statistical methods for rate and proportions will be used to assess binary outcomes, and standard methods for continuous data will be used for quantitative outcomes.

SECONDARY OUTCOMES:
Percentage of patients who experience hypoglycemia (defined as at least one blood glucose value less than 70) | Up to 2 years
  Standard statistical methods for rate and proportions will be used to assess binary outcomes, and standard methods for continuous data will be used for quantitative outcomes.
Percentage of patients who experience severe hypoglycemia (defined as at least one blood glucose value less than 40) | Up to 2 years
  Standard statistical methods for rate and proportions will be used to assess binary outcomes, and standard methods for continuous data will be used for quantitative outcomes.
Mean time to target range (100-140) | Up to 2 years
  Standard statistical methods for rate and proportions will be used to assess binary outcomes, and standard methods for continuous data will be used for quantitative outcomes.
Percentage of patients who experience hyperglycemia (defined as at least one blood glucose value greater than 200) 24 hours after initiation of infusion | 24 hours after initiation of infusion
  Standard statistical methods for rate and proportions will be used to assess binary outcomes, and standard methods for continuous data will be used for quantitative outcomes.
Percentage of patients who experience severe hyperglycemia (defined as at least one blood glucose value greater than 300) 24 hours after initiation of infusion | 24 hours after initiation of infusion
  Standard statistical methods for rate and proportions will be used to assess binary outcomes, and standard methods for continuous data will be used for quantitative outcomes.
Number of values greater than 200 or less than 70 per patient per day of treatment | Up to 2 years
  Standard statistical methods for rate and proportions will be used to assess binary outcomes, and standard methods for continuous data will be used for quantitative outcomes.
Glucose variability (defined as standard deviation of individual blood glucose values) | Up to 2 years
  Standard statistical methods for rate and proportions will be used to assess binary outcomes, and standard methods for continuous data will be used for quantitative outcomes.
Nursing satisfaction evaluated by the Glucose Monitoring Tool Trial Evaluation Form | Up to 2 years
  Standard statistical methods for rate and proportions will be used to assess binary outcomes, and standard methods for continuous data will be used for quantitative outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Merav Bar, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington